CLINICAL TRIAL: NCT02654977
Title: CLINICAL PROTOCOL to Investigate the Long-term Safety and Efficacy of Recombinant Human Leptin (METRELEPTIN) in Various Forms of Partial Lipodystrophy
Brief Title: CLINICAL PROTOCOL to Investigate the Long-term Safety and Efficacy of Metreleptin in Various Forms of Partial Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Professor, Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00093399
Record Dates: First submitted 2015-01-20; First posted 2016-01-13 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Familial Partial Lipodystrophy; Nonalcoholic Steatohepatitis; NAFLD
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Non-alcoholic Fatty Liver Disease | interventions — metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metreleptin (Experimental): Metreleptin open-label
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — MyaLept (Recombinant-methionyl Human Leptin (r-metHuLeptin) METRELEPTIN) subcutaneous injections
  Other Names: MyaLept

SUMMARY:
The study investigators' aim is to determine the long term safety and efficacy of Metreleptin (Myalept,) in promoting amelioration of metabolic abnormalities in patients with all forms of partial lipodystrophy. Patients will be offered this protocol under the following condition: Subjects have completed University of Michigan research protocol MB002-014 and have shown improved clinical benefit as judged by clinical criteria set forth in this protocol.

DETAILED DESCRIPTION:
Leptin is now an approved therapeutic in the form of Myalept in patients with generalized forms of lipodystrophy. However, it is still under investigation for patients with partial forms of the disease based on FDA decision on February 24, 2014. The study investigators have been carrying out a protocol in patients with partial lipodystrophy, specifically familial partial lipodystrophy. There have been a number of patients who have been treated under this protocol who are not covered by the currently approved label, but who have experienced significant clinical benefit.

This study allowed continued treatment of patients with partial forms of lipodystrophy who volunteered and completed treatment under the investigators' completed protocol (MB002-014) and who derived significant clinical benefit as judged by an amelioration of their hemoglobin A1c, triglyceride levels, and/or reduction in their baseline diabetes or lipid therapies that affect quality of life.

In this long-term study, there were three individuals whose data were excluded from final data analyses as explained in the results, however all participants were included in the presentation of baseline data as well as tabulated safety data.

ELIGIBILITY:
Inclusion Criteria:

* Previously completed study protocol:

  o CLINICAL PROTOCOL to investigate the efficacy of recombinant human leptin (METRELEPTIN) in nonalcoholic steatohepatitis (NASH) or nonalcoholic fatty liver disease (NAFLD) associated with lipodystrophy, MB002-014 (IRMBED: HUM00058708)
* Demonstrates clinical benefit as defined by meeting at least one of the following criteria upon completion of the above stated protocols:

  * Reduction of HbA1c ≥ 1.0% or,
  * Reduction of triglycerides ≥ 30% of baseline or,
  * Decrease in insulin requirements ≥ 40% or,
  * Reduction in total NASH score by ≥ 2 points,
  * Significant worsening of metabolic parameters after discontinuation of Metreleptin if discontinuation has been undertaken.
  * A health condition that appears to have significantly improved by metreleptin for which two independent health care providers make a request to prevent drug discontinuation. In addition, the PI has to document absence of contraindications for drug continuation (such as bone marrow suppression).
* Is male or female ≥ 5 years old at baseline.
* Is male, female not of childbearing potential, or meets all the following criteria if female of childbearing potential (including perimenopausal women who have had a menstrual period within one year):

  * Not breastfeeding
  * Negative pregnancy test result (human chorionic gonadotropin, beta subunit) at baseline (not applicable to hysterectomized females).
  * Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate when use consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire duration of metreleptin treatment.
* Has physician-confirmed lipodystrophy as defined by evidence of partial (limbs) loss of body fat outside the range of normal variation.
* If ≥ 18 years of age, is able to read, understand and sign the University of Michigan institutional review board (IRBMED) approved informed consent form (ICF), communicate with study physician and study team, understand and comply with protocol requirements.
* If < 18 and ≥ 7 years of age, is able to read, understand and sign the appropriate University of Michigan IRBMED approved assent form and has a parent or legal guardian that is able to read, understand and sign the ICF.
* If < 7 and ≥ 5 years of age or unable to read, the appropriate assent form must be explained to the child.
* If previously treated with thiazolidinediones or Vitamin E, stable dose of these medications for at least 3 months.

Exclusion Criteria:

* Presence of advanced liver disease (as evidenced by abnormal synthetic function, abnormal partial thromboplastin time or albumin).
* Evidence of other etiologies of viral hepatitis.
* Presence of clinically significant hematologic abnormalities (such as neutropenia and/or lymphadenopathy).
* Presence of HIV infection.
* Inability to give informed consent.
* Presence of end stage renal disease, any type of active cancer, or >class 2 congestive heart failure ((New York Heart Association Functional Classification System), based on medical history and physical examination.
* Has known allergies to E. coli-derived proteins or hypersensitivity to any component of metreleptin treatment.
* Any other condition in the opinion of the investigators that may impede successful data collection.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elif A Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metreleptin
Started | 11
Completed | 4
Not Completed | 7
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Metreleptin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Baseline triglyceride value [Median (Full Range); unit: mg/dL] — Minimum 10 hour fasting triglyceride value after completing 12 months of metreleptin in a prior study
  mg/dL | 204 [111 to 3047]
Baseline hemoglobin A1c value [Median (Full Range); unit: %] — Measured hemoglobin A1c value after completing 12 months of metreleptin in a prior study
  % | 8.4 [5.3 to 13.2]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fasting Triglyceride Levels
Description: Fasting triglyceride levels after 5 years on metreleptin, measured in mg/dL are compared to fasting triglyceride levels at baseline). The median percent increase (positive numbers) or decrease from baseline is shown, along with the full range.
Time Frame: 5 years on metreleptin or last observation carried forward
Population: Participants with immediate drop out, SAE withdrawal or death were excluded from analysis.
Measure: Median (Full Range); unit: percentage of change from baseline
Arm/Group | Metreleptin
Number analyzed (Participants) | 8
percentage of change from baseline | 55.76 [-66.79 to 203.80]

2. Secondary Outcome: Percent Change in Hemoglobin A1c Levels
Description: Fasting hemoglobin A1c levels after 5 years on metreleptin, measured in % are compared to fasting Hemoglobin levels at baseline). Thus, for example, a change from 10% to 5% would be a -50% change (or 50% decrease). The median percent increase (positive numbers) or decrease from baseline is shown, along with the full range.
Time Frame: 5 years on metreleptin or last observation carried forward
Population: Percent change in hemoglobin A1c levels (hemoglobin A1c levels are measured in %) Participants with immediate drop out, SAE withdrawal or death were excluded from analysis.
Measure: Median (Full Range); unit: percentage of change from baseline
Arm/Group | Metreleptin
Number analyzed (Participants) | 8
percentage of change from baseline | 2.55 [-27.52 to 25.00]

ADVERSE EVENTS:
Time Frame: 5 years (from baseline visit to year 5 study visit or date of study participant early termination)
Arm/Group | Metreleptin
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin (N=11)
anterior cervical discectomy (Surgical and medical procedures) | 1 (1)
labia majora dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
onset of type 1 diabetes (Endocrine disorders) | 1 (1)
Onset of hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
diabetic ketoacidosis (Endocrine disorders) | 1 (4)
hypokalemia (Endocrine disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (2)
pancreatitis (Endocrine disorders) | 1 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
metreleptin neutralizing antibodies (Immune system disorders) | 1 (1)
acute hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
left shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
nonepilogenic seizures (Nervous system disorders) | 1 (1)
clinical sepsis (Infections and infestations) | 1 (1)
splenic flexure colitis fluid collection (Gastrointestinal disorders) | 1 (1)
multiple rib fractures (Musculoskeletal and connective tissue disorders) | 1 (1)
splenic laceration (Gastrointestinal disorders) | 1 (1)
uterine bleeding (Reproductive system and breast disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2)
dizziness (Nervous system disorders) | 1 (1)
chest pain with elevated troponin (Cardiac disorders) | 1 (2)
atrial flutter (Cardiac disorders) | 1 (1)
sudden cardiac death (Cardiac disorders) | 1 (1) — as listed in All Cause Mortality
chronic heart failure exacerbation (Cardiac disorders) | 1 (1)
cholecystitis (Gastrointestinal disorders) | 1 (1)
esophageal spasms (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin (N=11)
worsening of chronic back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
hyperesthesia (Nervous system disorders) | 1 (1)
sinus infection (Infections and infestations) | 1 (1)
extremity weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
cold (Infections and infestations) | 3 (3)
weight loss (Endocrine disorders) | 1 (1)
elevated liver function tests (Metabolism and nutrition disorders) | 1 (1)
acid reflux (Gastrointestinal disorders) | 1 (1)
cellutitus (Infections and infestations) | 2 (5)
kidney stone (Renal and urinary disorders) | 1 (1)
strep throat (Infections and infestations) | 1 (1)
reticular rash (Skin and subcutaneous tissue disorders) | 2 (2)
urinary tract infection (Infections and infestations) | 3 (5)
hypoglycemia (Endocrine disorders) | 2 (4)
nausea (Gastrointestinal disorders) | 1 (2)
headache (Nervous system disorders) | 1 (1)
worsening vitamin D deficiency (Endocrine disorders) | 1 (1)
worsening imbalance (Nervous system disorders) | 1 (1)
worsening diabetes (Endocrine disorders) | 1 (1)
worsening weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 3 (3)
vomiting (Gastrointestinal disorders) | 1 (1)
bronchitis (Infections and infestations) | 2 (2)
increase in appetite (Endocrine disorders) | 1 (1)
cardiac chest pain (Cardiac disorders) | 1 (1)
lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
elevated blood platelets (Blood and lymphatic system disorders) | 2 (2)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
vaginal spotting (Reproductive system and breast disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
vaginal yeast infection (Infections and infestations) | 1 (3)
elevated low density cholesterol (Metabolism and nutrition disorders) | 1 (1)
worsening of restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
low blood iron level (Endocrine disorders) | 1 (1)
infected tooth (Infections and infestations) | 1 (1)
kidney infection (Infections and infestations) | 1 (1)
thyroid nodules (Metabolism and nutrition disorders) | 1 (1)
intermittent suicidal ideation (Psychiatric disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 3 (3)
increased blood protein levels (Blood and lymphatic system disorders) | 1 (1)
worsening depression (Psychiatric disorders) | 3 (3)
right wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1)
right wrist numbness (Musculoskeletal and connective tissue disorders) | 1 (1)
lower right leg numbness (Musculoskeletal and connective tissue disorders) | 1 (1)
irregular periods (Reproductive system and breast disorders) | 1 (1)
worsening of fecal incontinence (Gastrointestinal disorders) | 1 (1)
retinopathy lesion (Eye disorders) | 1 (1)
frozen shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
abnormal stress test (Cardiac disorders) | 1 (1)
viral illness (Infections and infestations) | 1 (1)
worsening cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
increased creatitine levels (Endocrine disorders) | 1 (1)
blocked parotid gland (Infections and infestations) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
ostearthritis dissicans (Musculoskeletal and connective tissue disorders) | 1 (1)
worsening anxiety (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Definitive conclusions cannot be drawn from sample sizes as small as the four individuals who completed the trial period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT02654977/Prot_000.pdf